CLINICAL TRIAL: NCT06529055
Title: Effects of Oral Nicotine and Caffeine Pouches on Anaerobic Performance, Autonomic Function, Cognition, and Behavior
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Responsible Party: Principal Investigator, Austin Graybeal, Assistant Professor, University of Southern Mississippi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-0285
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Fatigue; Muscle, Heart; Fatigue, Mental
MeSH Terms: conditions — Fatigue; Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oral Nicotine Pouches (Experimental): Single dose 3mg oral nicotine pouch
  Interventions: Other: Oral Pouch - Nicotine
- Oral Caffeine Pouches (Experimental): Single dose 100mg oral caffeine pouch
  Interventions: Other: Oral Pouch - Caffeine
- Combination of oral nicotine and caffeine pouches (Experimental): Single simultaneous doses of a 3mg oral nicotine pouch and a 100mg oral caffeine pouch
  Interventions: Other: Oral Pouch - Nicotine; Other: Oral Pouch - Caffeine
- Placebo (Placebo Comparator): Flavor, color, and appearance matched placebo
  Interventions: Other: Oral Pouch - Placebo

INTERVENTIONS:
Other: Oral Pouch - Nicotine — Ingestion of a randomized oral nicotine pouch
  Arms: Combination of oral nicotine and caffeine pouches; Oral Nicotine Pouches
Other: Oral Pouch - Caffeine — Ingestion of a randomized oral caffeine pouch
  Arms: Combination of oral nicotine and caffeine pouches; Oral Caffeine Pouches
Other: Oral Pouch - Placebo — Ingestion of a randomized oral placebo pouch
  Arms: Placebo

SUMMARY:
The goal of this randomized placebo controlled crossover trial is to determine effects of oral nicotine and caffeine pouches on anaerobic performance, autonomic function, cognition, and behavior in adult non-obese adult male volunteers between ages 21 and 40.

Accordingly, the primary aims of the study are to determine the effects of acute oral nicotine pouches, oral caffeine pouches, or both, on measures of

* anaerobic performance
* cognition
* cardiovascular and autonomic function
* appetite and food intake.

Researchers will compare oral nicotine pouches, oral caffeine pouches, both oral nicotine and caffeine pouches, and a flavor and color matched placebo to see if how they differentially affect measurements of

* physical performance,
* cognition,
* cardiovascular and autonomic function
* appetite and food intake.

On four separate occasions, participants will be asked to place the oral pouches in their mouth and complete several anerobic cycling, cognitive, and balance tests while blood and salivary biomarkers, subjective appetite ratings, and cardiovascular and autonomic function measurements are collected. After each trial, participants will complete a 24-hr food record.

ELIGIBILITY:
Inclusion Criteria:

* Being 21 to 40 years of age
* Being biologically male
* Having a body mass index (BMI) of < 30 kilograms/meter-squared
* Participating in moderate/vigorous exercise for at least 150 minutes/week over the last month

Exclusion Criteria:

* individuals who are younger than 21 or older than 40
* missing any limbs or part of a limb
* having any neuromuscular/musculoskeletal injury or impairment that would prevent performing any exercise/functional measures for this study
* having a pacemaker or any other electrical implant
* a diagnosis (defined as the presence of disease of or using medication to treat the disease) of heart failure, cardiomyopathy (dilated or hypertrophic), valvular disease, type I or type II diabetes
* taking insulin injections
* any history of severe or mild traumatic brain injury within the last two years
* kidney, liver, thyroid, or heart disease
* treated or untreated American Heart Association stage 2 hypertension (>140 millimeters of mercury / > 90 millimeters of mercury)
* any diagnosed neurological or neurodegenerative diseases
* having donated blood or plasma in the last 20 days prior to blood collection procedures
* taking any supplements/medications that may interfere with the results of the study
* any surgeries that would impact swallowing and/or digestion
* currently smoking, vaping, using e-cigarettes, or using any other combustible/smokeless tobacco products
* using smokeless tobacco-free nicotine products on more than 2 days/week
* daily caffeine use of more than 250 milligrams/day or use of any oral caffeine pouches
* have allergies or are regularly taking medications that would impact this study and/or negatively interact with caffeine or nicotine.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wingate Anaerobic Cycling Test | Baseline, 15, 16, 19, 20, 23, 24, 27, 28, 31, 32, and 60 minutes post-ingestion
  Changes in anaerobic cycling power output
Concentration of blood lactate | Baseline, 25, 32 minutes post-ingestion
  Changes in blood lactate concentration from capillary blood
Concentration of salivary cortisol | Baseline, 15, 25, 32 minutes post-ingestion
  Changes in salivary cortisol concentration from saliva
Concentration of salivary interleukin-6 | Baseline, 15, 25, 32 minutes post-ingestion
  Changes in interleukin-6 concentration from saliva
Salivary catecholamine concentration | Baseline, 15, 27, 40 minutes post-ingestion
  Changes in salivary catecholamine concentration from saliva
Profile of Mood States | Baseline, 15, 32 minutes post-ingestion
  Changes in Profile of Mood States scores (Score range: 0-60)
Balance | Baseline, 15, 32 minutes post-ingestion
  Changes in standing postural sway
Ratings of perceived exertion | Baseline, 15, 16, 19, 20, 23, 24, 27, 28, 31, 32, and 60 minutes post-ingestion
  Changes in ratings of perceived exertion (Scale range: 6-20 - lower ratings means less effort))
Hunger - Visual Digital Analog Scale (0-100) | Baseline, 15, 25, 32 minutes post-ingestion
  Changes in subjective ratings of hunger
Desire to eat - Visual Digital Analog Scale (0-100) | Baseline, 15, 25, 32, 60 minutes post-ingestion
  Changes in subjective ratings of desire to eat
Prospective Consumption of Food - Visual Digital Analog Scale (0-100) | Baseline, 15, 25, 32, 60 minutes post-ingestion
  Changes in subjective ratings of prospective consumption of food
Fullness - Visual Digital Analog Scale (0-100) | Baseline, 15, 25, 32, 60 minutes post-ingestion
  Changes in subjective ratings of fullness
Food Intake - Digital 24-hour food record | 24 hours following the end of each visit
  Consumption of food and beverage after study visit
Blood Pressure | Baseline, 15, 19, 23, 27, 31, and 60 minutes post-ingestion
  Absolute brachial blood pressure values (systolic and diastolic) and relative changes from baseline.
Heart Rate | Baseline, 15, 19, 23, 27, 31, and 60 minutes post-ingestion
  Absolute heart rate values and relative changes from baseline.
Trail Making Test - Digital Cognitive Function Test | Baseline, 15, 32 minutes post-ingestion
  Changes in trail making test scores
Sustained Attention Test - Digital Cognitive Function Test | Baseline, 15, 32 minutes post-ingestion
  Changes in sustained attention test scores
Visual Working Memory Span Test - Digital Cognitive Function Test | Baseline, 15, 32 minutes post-ingestion
  Changes in visual working memory span test scores
Stroop Test - Digital Cognitive Function Test | Baseline, 15, 32 minutes post-ingestion
  Changes in Stroop test scores
Deary-Liewald Test - Digital Cognitive Function Test | Baseline, 15, 32 minutes post-ingestion
  Changes in Deary-Liewald test scores
Cerebral Blood flow | Baseline, 15, 19, 23, 27, and 31 minutes post-ingestion
  Doppler ultrasound derived blood flow in the carotid artery

SECONDARY OUTCOMES:
Blood Glucose Concentration | Baseline, 15, 25, 32 minutes post-ingestion
  Changes in blood glucose concentration from capillary blood
Salivary insulin concentration | Baseline, 15, 25, and 32 minutes post-ingestion
  Changes in salivary insulin concentration from saliva
Prefrontal Cortex Oxygenation | Baseline, 15, 19, 23, 27, and 31 minutes post-ingestion
  Near-infrared spectroscopy
Peripheral Vascular Conductance | Baseline, 15, 19, 23, 27, and 31 minutes post-ingestion
  Blood flow in the brachial artery normalized to blood pressure (mL/min/mmHg)
Electromyography | Baseline, 15, 16, 19, 20, 23, 24, 27, 28, 31, and 32 minutes post-ingestion
  Electromyographic reading of muscle activity of the active muscles (glutes, hamstrings, quadriceps, and calves)
Peripheral Blood Flow | Baseline, 15, 19, 23, 27, and 31 minutes post-ingestion
  Doppler ultrasound derived blood flow in the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Austin J Graybeal, PhD, Principal Investigator — University of Southern Mississippi
Locations (1):
- University of Southern Mississippi - School of Kinesiology and Nutrition, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No